CLINICAL TRIAL: NCT06113471
Title: A Phase 3, Randomized, Double-Blind, 52-Week, Placebo-Controlled, Efficacy and Safety Study of Povorcitinib in Participants With Nonsegmental Vitiligo
Brief Title: A Study to Evaluate Efficacy and Safety of Povorcitinib in Participants With Nonsegmental Vitiligo (STOP-V2)
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Incyte Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: INCB54707-304; 2023-506011-18-00 (Registry Identifier: EU CT Number)
Record Dates: First submitted 2023-10-27; First posted 2023-11-02 (Actual); Last update posted 2026-02-03 (Actual); Status verified 2026-01

CONDITIONS: NonSegmental Vitiligo

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Experimental: Povorcitinib Dose A (Experimental): Participants will receive Povorcitinib Dose A for 52 weeks, followed by Povorcitinib Dose A for 52 weeks.
  Interventions: Drug: Povorcitinib
- Placebo (Placebo Comparator): Participants will receive Placebo for 52 weeks, followed by Povorcitinib Dose A for 52 weeks.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Povorcitinib — Oral, Tablet
  Other Names: INCB054707
  Arms: Experimental: Povorcitinib Dose A
Drug: Placebo — Oral, Tablet
  Arms: Placebo

SUMMARY:
This study is being conducted to determine the efficacy and safety of povorcitinib in participants with nonsegmental vitiligo.

ELIGIBILITY:
Inclusion Criteria:

* Aged ≥ 18 years.
* Clinical diagnosis of nonsegmental vitiligo and meet the following:

  * T-BSA ≥ 5%
  * T-VASI score ≥ 4
  * F-BSA ≥ 0.5%
  * F-VASI score ≥ 0.5
* Agreement to discontinue all agents and procedures used to treat vitiligo from screening through the final safety follow-up visit.
* Willingness to avoid pregnancy or fathering children.

Exclusion Criteria:

* Other forms of vitiligo or skin depigmentation disorders.
* Clinically significant abnormal TSH or free T4 at screening.
* Use of laser or phototherapy within 8 weeks and dihydroxyacetone within 4 weeks prior to Day 1.
* Current or past use of the depigmenting agent monobenzyl ether of hydroquinone including Benoquin®.
* History of melanocyte-keratinocyte transplantation procedure or other surgical treatment for vitiligo.
* Spontaneous and significant repigmentation within 6 months prior to screening.
* Women who are pregnant, considering pregnancy, or breast feeding.
* Medical history including thrombocytopenia, coagulopathy or platelet dysfunction; venous and arterial thrombosis, deep vein thrombosis, pulmonary embolism, stroke, moderate to severe heart failure, cerebrovascular accident, myocardial infarction, or other significant cardiovascular diseases; Q-wave interval abnormalities; disseminated herpes zoster or recurrent dermatomal herpes zoster; disseminated herpes simplex; chronic/recurrent infections; malignancies.
* Evidence of infection with TB, HBV, HCV or HIV.
* History of failure to JAK inhibitor treatment of any inflammatory disease.
* Laboratory values outside of the protocol-defined ranges.

Other protocol-defined Inclusion/Exclusion Criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 450 (Actual)
Dates: Start 2023-11-27 (Actual); Primary Completion 2026-03-17 (Estimated); Study Completion 2027-03-16 (Estimated)

PRIMARY OUTCOMES:
Proportion of Participants Achieving a ≥ 75% Improvement From Baseline in the Facial Vitiligo Area Scoring Index (F-VASI75) | Week 52
  ≥75% improvement in facial Vitiligo Area Scoring Index.

SECONDARY OUTCOMES:
Percentage change from Baseline in Total Body Vitiligo Area Scoring Index (T-VASI) | Week 52
  Percentage change from Baseline in total body Vitiligo Area Scoring Index.
Proportion of Participants Achieving a ≥ 50% Improvement From Baseline in the Total Body Vitiligo Area Scoring Index (T-VASI50) | Week 52
  ≥50% improvement in total body Vitiligo Area Scoring Index.
Proportion of Participants Achieving a ≥ 75% Improvement From Baseline in the Total Body Vitiligo Area Scoring Index (T-VASI75) | Week 52
  ≥75% improvement in total body Vitiligo Area Scoring Index.
Proportion of participants achieving a Vitiligo Noticeability Scale Score (VNS) of 4 or 5 | Week 52 and Week 104
  VNS is a participant reported outcome measure on a scale of 1-5, 1- more noticeable, 4 - a lot less noticeable, and 5- no longer noticeable.
Number of participants with Treatment-emergent Adverse Events (TEAEs) | Up to Week 104 and 30 days
  Defined as adverse events reported for the first time or worsening of a pre-existing event after first dose of study drug.
Proportion of Participants Achieving Facial Vitiligo Area Scoring Index (F-VASI50) | Week 52 and Week 104
  ≥50% improvement in facial Vitiligo Area Scoring Index.
Proportion of Participants Achieving Facial Vitiligo Area Scoring Index (F-VASI75) | Week 104
  ≥75% improvement in facial Vitiligo Area Scoring Index.
Proportion of Participants Achieving Facial Vitiligo Area Scoring Index (F-VAS190) | Week 52 and Week 104
  ≥90% improvement in facial Vitiligo Area Scoring Index.
Proportion of Participants Achieving Total Body Vitiligo Area Scoring Index (T-VASI50) | Week 104
  ≥50% improvement in total body Vitiligo Area Scoring Index.
Proportion of Participants Achieving Total Body Vitiligo Area Scoring Index (T-VASI75) | Week 104
  ≥75% improvement in total body Vitiligo Area Scoring Index.
Proportion of Participants Achieving Total Body Vitiligo Area Scoring Index (T-VASI90) | Week 52 and Week 104
  ≥90% improvement in total body Vitiligo Area Scoring Index.
Proportion of participants achieving an Facial Static Investigator Global Assessment (FSIGA) of 0 or 1 | Week 52 and Week 104
  Global score of vitiligo severity for the face. Scores range from 0 (clear) to 5 (severe vitiligo).
Proportion of participants in each Facial Static Investigator Global Assessment (FSIGA) category | Week 52 and Week 104
  Global score of vitiligo severity for the face. Scores range from 0 (clear) to 5 (severe vitiligo).
Proportion of participants achieving a Static Investigator Global Assessment (SIGA) of 0 (clear) or 1 (almost clear) | Week 52 and Week 104
  Global score of vitiligo severity for the entire body. Scores range from 0 (clear) to 5 (severe vitiligo).
Proportion of participants in each Static Investigator Global Assessment (SIGA) category | Week 52 and Week 104
  Global score of vitiligo severity for the entire body. Scores range from 0 (clear) to 5 (severe vitiligo).
Proportion of participants who report Facial Patient Global Impression of Change-Vitiligo (F-PaGIC-V) of 1 or 2 | Week 52 and Week 104
  F-PaGIC-V is an assessment of improvement of vitiligo on the face by the participant. It is a 7-point scale ((1) Very much improved, (2) Much improved, (3) Minimally improved, (4) No change, (5) Minimally worse, (6) Much worse, or (7) Very much worse).
Proportion of participants in each Facial Patient Global Impression of Change-Vitiligo (F-PaGIC-V) category | Week 52 and Week 104
  F-PaGIC-V is an assessment of improvement of vitiligo on the face by the participant. It is a 7-point scale ((1) Very much improved, (2) Much improved, (3) Minimally improved, (4) No change, (5) Minimally worse, (6) Much worse, or (7) Very much worse).
Proportion of participants who report Total Body Patient Global Impression of Change-Vitiligo (T-PaGIC-V) of 1 or 2 | Week 52 and Week 104
  T-PaGIC-V is an assessment of improvement of vitiligo on the total body by the participant. It is a 7-point scale ((1) Very much improved, (2) Much improved, (3) Minimally improved, (4) No change, (5) Minimally worse, (6) Much worse, or (7) Very much worse).
Proportion of participants in each Total Body Patient Global Impression of Change-Vitiligo (T-PaGIC-V) category | Week 52 and Week 104
  T-PaGIC-V is an assessment of improvement of vitiligo on the total body by the participant. It is a 7-point scale ((1) Very much improved, (2) Much improved, (3) Minimally improved, (4) No change, (5) Minimally worse, (6) Much worse, or (7) Very much worse).
Proportion of participants in each category for the color-matching question | Week 52 and Week 104
  Participants will answer how well the color of the treated skin matches the normal skin on a scale of 1-5, 1 being excellent to 5 being very poor.
Change from baseline in the Vitiligo-Specific Quality of Life (VitiQoL) | Week 52 and Week 104
  VitiQoL is a 15-item QoL assessment that asks participants to rate various aspects of their condition during the past month using a 7-point scale ("Not at all" to "All of the time").
Change from baseline in the Hospital Anxiety and Depression Scale (HADS) subscales | Week 52 and Week 104
  HADS is a 14-item questionnaire that assesses the levels of anxiety and depression that a participant is currently experiencing. There are 7 questions each for measuring anxiety and for measuring depression, with 4 possible responses to each question (responses are scored as 0, 1, 2, or 3).

CONTACTS AND LOCATIONS:
Overall Officials: Incyte Medical Monitor, Study Director — Incyte Corporation
Locations (86):
- United States (33):
  - University of Alabama At Birmingham Hospital-Whitaker Clinic, Birmingham, Alabama
  - C2 Research Center, Llc, Montgomery, Alabama
  - First Oc Dermatology Research Inc, Fountain Valley, California
  - Center For Dermatology Clinical Research, Inc, Fremont, California
  - Marvel Clinical Research Llc, Huntington Beach, California
  - Vitiligo & Pigmentation Institute of Southern California, Los Angeles, California
  - Dermatology Research Associates, Los Angeles, California
  - Clinical Trials Research Institute, Thousand Oaks, California
  - Skin Care Research, Llc, Boca Raton, Florida
  - Total Vein and Skin Llc, Boynton Beach, Florida
  - Driven Research Llc, Coral Gables, Florida
  - Florida Academic Centers Research and Education Llc, Coral Gables, Florida
  - Pediatric Skin Research Llc, Coral Gables, Florida
  - Metabolic Research Institute Inc, West Palm Beach, Florida
  - Dermatology and Surgery Specialists of North Atlanta, Marietta, Georgia
  - Advanced Medical Research Pc, Sandy Springs, Georgia
  - Dundee Dermatology, West Dundee, Illinois
  - Indiana University School of Medicine Iusm Indianapolis, Indianapolis, Indiana
  - Delricht Research, Baton Rouge, Louisiana
  - Callender Dermatology and Cosmetic Center, Glenn Dale, Maryland
  - Aesthetic and Dermatology Center, Rockville, Maryland
  - Henry Ford Health System, Detroit, Michigan
  - Allcutis Research, Llc, Portsmouth, New Hampshire
  - Weill Cornell Medical College, New York, New York
  - Remington-Davis Clinical Research, Columbus, Ohio
  - Oregon Medical Research Center, Pc, Portland, Oregon
  - Dermatology Treatment and Research Center, Dallas, Texas
  - Heights Dermatology and Aesthetic Center, Houston, Texas
  - University of Texas, Md Anderson Cancer, Houston, Texas
  - Innovative Dermatology: Legacy Medical Village, Plano, Texas
  - Texas Dermatology and Laser Specialists, San Antonio, Texas
  - Dermatology Clinical Research Center of San Antonio, San Antonio, Texas
  - Premier Clinical Research, Spokane, Washington
- Bulgaria (5):
  - Medical Center Asklepii Ood, Dupnitsa
  - Medical Center Unimed Eood, Sliven
  - Ambulatory For Specialized Medical Care - Individual Practice For Specialized Medical Care - Skin An, Sofia
  - Aleksandrovska University Hospital, Sofia
  - 28 Diagnostic and Consultative Center, Sofia
- Canada (6):
  - British Columbia'S Centre For Dermatologic Science - the Skin Care Centre, Vancouver, British Columbia
  - Lynderm Research Inc, Markham, Ontario
  - DERMEDGE, Mississauga, Ontario
  - Toronto Research Centre, Toronto, Ontario
  - Research Toronto, Toronto, Ontario
  - Centre de Recherche Dermatologique de Quebec, Québec, Quebec
- France (5):
  - Chru Morvan/Chu Brest Hopital Morvan, Brest
  - Centre Hospitalier - Le Mans, Le Mans
  - Cabinet Medical- Chemin de Paradis, Martigues
  - Centre Hospitalier Universitaire de Nice,Hopital L Archet, Nice
  - Hopital Charles Nicolle, Rouen
- Germany (6):
  - Fachklinik Bad Bentheim, Bad Bentheim
  - Charite Universitaetsmedizin Berlin - Campus Charite Mitte, Berlin
  - University Hospital Carl Gustav Carus, Dresden
  - Universitaetsklinikum Hamburg-Eppendorf, Hamburg
  - Dermatologische Gemeinschaftspraxis, Mahlow
  - Universitaetsklinikum Muenster, Münster
- Hungary (3):
  - Orvostudomanyi Kutato Es Fejleszto Kft, Debrecen
  - Debreceni Egyetem, Debrecen
  - Markusovszky Teaching Hospital, Szombathely
- Italy (5):
  - Asst Degli Spedali Civili Di Brescia, Brescia
  - Azienda Policlinico Vittorio Emanuele, Catania
  - Fondazione Irccs Ca Granda Ospedale Maggiore, Milan
  - Fondazione Policlinico Universitario Agostino Gemelli Irccs, Rome
  - Irccs Istituto Clinico Humanitas, Rozzano
- Poland (18):
  - Synexus Polska Sp. Z O.O. Oddzial W Gdansku, Gdansk
  - Synexus Gdynia, Gdynia
  - Provita Sp.Zo.O. Centrum Medyczne Angelius, Katowice
  - Pro Familia Altera Sp. Z O.O., Katowice
  - Prywatny Gabinet Dermatologiczny Elzbieta Klujszo, Kielce
  - Niepubliczny Zaklad Opieki Zdrowotnej Dermed Centrum Medyczne Sp. Z O.O., Lodz
  - Dermoklinika Centrum Medyczne S.C., M. Kierstan, J. Narbutt, A. Lesiak, Lodz
  - Velocity Clinical Research, Skierniewice, Skierniewice
  - Laser Clinic, Szczecin
  - Twoja Przychodnia - Szczecinskie Centrum Medyczne, Szczecin
  - Alergo-Med Specjalistyczna Przychodnia Lekarska Sp. Z O.O., Tarnów
  - Centrum Medyczne Evimed, Warsaw
  - Royalderm Agnieszka Nawrocka, Warsaw
  - Klinika Ambroziak Sp. Z O.O., Warsaw
  - Futuremeds Targowek Centrum Medyczne Amed Warszawa Targowek, Wrocaw
  - Synexus Polska Sp. Z O.O. Oddzial We Wroclawiu, Wroclaw
  - Dermmedica Sp. Z O.O., Wroclaw
  - Centrum Medyczne Oporow, Wroclaw
- United Kingdom (5):
  - Ipswich Hospital, East Suffolk and North Essex Nhs Foundation Trust, Ipswich
  - University Hospitals of Leicester-Leicester Royal Infirmary (Lri), Leicester
  - Whipps Cross University Hospital - Barts Health Nhs Trust, London
  - Nottingham University Hospitals - Treatment Center, Nottingham
  - Royal Wolverhampton Nhs Trust, Walsall

IPD SHARING:
Plan to Share IPD: Yes
Incyte shares data with qualified external researchers after a research proposal is submitted. These requests are reviewed and approved by a review panel on the basis of scientific merit. All data provided is anonymized to respect the privacy of patients who have participated in the trial in line with applicable laws and regulations.
  The trial data availability is according to the criteria and process described on https://www.incyte.com/our-company/compliance-and-transparency
Supporting Information: Study Protocol, SAP
Time Frame: Data will be shared after the primary publication or 2 years after the study has ended for market authorized products and indications.
Access Criteria: Data from eligible studies will be shared with qualified researchers according to the criteria and process described in the Data Sharing section of the www.incyteclinicaltrials.com website. For approved requests, the researchers will be granted access to anonymized data under the terms of a data sharing agreement.
URL: https://www.incyte.com/our-company/compliance-and-transparency

REFERENCES:
- See also: A study to Evaluate Efficacy and Safety of Povorcitinib in Participants With Nonsegmental Vitiligo (STOP-V2) — https://www.incyteclinicaltrials.com/study/?id=INCB54707-304&SearchTerm=INCB54707-304&Latitude=&Longitude=&LocationName=&conditions=&Status=&phases=&AgeRanges=&gender=&StudyTypes=&AttachmentTypes=&MileRadius=100&PageIndex=0&PageSize=10&SortField=&SortOrder=&hasResults=